CLINICAL TRIAL: NCT04836000
Title: Effectiveness of Low-level Laser Therapy in Patients With Arthroscopic Rotator Cuff Repair
Brief Title: Effectiveness of Low-level Laser Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner Karartı, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021100
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Tears; Rehabilitation; Rotator Cuff Injuries
Keywords: Laser Therapy; Low-Level; Biostimulation; Phototherapy; Rotator Cuff Injuries; Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): In addition to the conservative treatment of the control group, low-level laser therapy (turned off) will be applied for 6 weeks. In the placebo group, laser instrument will be applied in the same way but the device will be turned off during treatment sessions.
  Interventions: Other: In addition to the conservative treatment, Low-level laser therapy (turned off)
- Experimental Group (Experimental): In addition to the conservative treatment of the control group, low-level laser therapy will be applied for 6 weeks.
  Interventions: Other: In addition to the conservative treatment, Low-level laser therapy
- Control Group (Active Comparator): For 6 weeks, all three groups will receive five sessions per week of a protocolised treatment based on therapeutic exercises, analgesic electrotherapy and cryotherapy.
  Interventions: Other: Conservative treatment solely

INTERVENTIONS:
Other: In addition to the conservative treatment, Low-level laser therapy — For Experimental Group A Gallium-aluminum-arsenide (Ga-Al-As) diode laser instrument (Roland Serie, Elettronica Pagani, Paderno, Italy, Mod IR 27/1) will be used (wavelength 904 nm, 5500 Hz frequency, 27 W maximum power output per pulse, 13.2 mW average power, 0.8-cm2 spot size, 1.6 J of total energy will be delivered per point at each session at a power density of 16.5 mW/cm2, and the cumulative energy per point for all sessions was 16 J).
  Ga-Al-As laser therapy will be applied to experimental group patients two times per week for 6 weeks in 10-min sessions. LLLT will be applied over the tuberculum majus and minus, the anterior and posterior faces of the capsule, and the subacromial regions. Each point will be treated for 120 sec. The head of the instrument will be held perpendicular to the body surface and in skin contact without pressure.
  Arms: Experimental Group
Other: In addition to the conservative treatment, Low-level laser therapy (turned off) — For Placebo Group In the placebo group, laser instrument will be applied in the same way but the device will be turned off during treatment sessions. Patients and physiotherapist will be asked to use protective eyeglasses during therapy for safety.
  Arms: Placebo Group
Other: Conservative treatment solely — For Control Group All patients using an immobilization bandage up to post-operative 6th week will receive the standardized 6-week supervised rehabilitation program advocated by the same physiotherapist (CK), 7 years of experience in the clinical treatment of rotator cuff tear, after the baseline assessment. Composed of 30 treatment sessions (five days/week) of 45 to 60 minutes, the rehabilitation program will be provided individually to all participants. Physiotherapy sessions will be devoted to strength, mobilizations, stretching, perturbation, and sensorimotor training using motor control exercises, hence, to restore adequate shoulder neuromuscular control. The treatment program will also be included patient education.
  Arms: Control Group

SUMMARY:
During rotator cuff tear healing stages, there are complex interactions between a variety of tissue growth factors and cells, ultimately resulting in tissue that is markedly different from that of normal, uninjured tendon. Hence, there is a strong drive to investigate the role of potential therapies in the form of biological augments that may restore the pathologic tissue to a near normal physiological state. In this context, low-level laser therapy (LLLT) may be an effective choice in the treatment of nonoperative small and medium-sized rotator cuff tears (RCT). To the best of our knowledge, there is no randomized controlled study investigating the effects of the LLLT in patients with a arthroscopic rotator cuff repair (ARCR). Therefore, the aim of the current study is to investigate all the possible effects of the LLLT in terms of functional status, pain-free mobility, and quality-of-life.

DETAILED DESCRIPTION:
Recently, there is a increasing evidence that the addition of low-level laser therapy (LLLT) to treatment program of shoulder problems plays an important role in stimulation of healing, augmenting tissue repair, relief of pain and inflammation, and restoration of function. LLLT, phototherapy or photobiomodulation refers to the use of photons at a non-thermal irradiance to alter biological activity. The basic biological mechanism behind the effects of LLLT is thought to be through absorption of red and near infrared light by mitochondrial chromophores, in particular cytochrome c oxidase (CCO) which is contained in the respiratory chain located within the mitochondria, and perhaps also by photoacceptors in the plasma membrane of cells. It is hypothesized that this absorption of light energy may cause photodissociation of inhibitory nitric oxide from CCO9 leading to enhancement of enzyme activity, electron transport, mitochondrial respiration and adenosine triphosphate (ATP) production. In turn, LLLT alters the cellular redox state which induces the activation of numerous intracellular signaling pathways, and alters the affinity of transcription factors concerned with cell proliferation, survival, tissue repair and regeneration.

During rotator cuff tear healing stages, there are complex interactions between a variety of tissue growth factors and cells, ultimately resulting in tissue that is markedly different from that of normal, uninjured tendon. Hence, there is a strong drive to investigate the role of potential therapies in the form of biological augments that may restore the pathologic tissue to a near normal physiological state. In this context, LLLT may be an effective choice in the treatment of nonoperative small and medium-sized rotator cuff tears (RCT). o the best of our knowledge, there is no randomized controlled study investigating the effects of the LLLT in patients with a arthroscopic rotator cuff repair (ARCR). Therefore, the aim of the current study is to investigate all the possible effects of the LLLT in terms of functional status, pain-free mobility, and quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* being 18-65 years old
* being diagnosed with a rotator cuff tear not exceeding 3 cm based on magnetic resonance imaging and clinical continuity tests
* history of arthroscopic rotator cuff tear
* using a velpeau bandage up to post-operative 6th week
* compliance to range of motion (ROM) exercises including pendulum exercises, passive flexion and abduction stretching, and active cervical movements
* volunteering to participate in the study.

Exclusion Criteria:

* Patients with diabetes mellitus
* neurological problems
* cervical disc herniation
* visual, verbal, and/or cognitive defects
* systemic inflammatory problems
* trauma
* contraindications for mobilization
* former shoulder fractures and surgery
* a history of adhesive capsulitis
* traumatic shoulder instability
* patients who were in ≥stage 3 on the Goutallier system
* those who received a corticosteroid injection on the affected side within 6 weeks prior to diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Constant-Murley score (Functional Outcome) | 6 weeks
  It assesses four aspects related to shoulder pathology; two subjective: pain and activities of daily living (ADL) and two objective: range of motion (ROM) and strength. The subjective components can receive up to 35 points and the objective 65, resulting in a possible maximum total score of 100 points (best function). Pain and ADL are answered by the patient; ROM and strength require a physical evaluation and are answered by the orthopaedic surgeon or the physiotherapist

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff index (Functional Outcome and Quality of life) | 6 weeks
  It is a self-administering health questionnaire. It has 21 items, exploring 5 different domains: Physical symptoms, Sports and recreation, Work, Social function, Emotions. Each question uses a visual analogue scale (VAS) - which is a straight line, representing a 100-point scale, ranging from 0-100. The maximum score is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all. To make the final score more clinically friendly, some minor math is involved. The score can be reported as a percentage by subtracting the total from 2100, dividing by 2100, and multiplying by 100. This will give you an overall percentage. Total final WORC scores can, therefore, range from 0% ( lowest functional status level) to 100% (the highest functional status).
Pain-free mobility of the shoulder | 6 weeks
  Pain-free flexion and abduction will be assessed with universal goniometer.
EQ-5D-5L (quality-of-life) | 6 weeks
  The 5-level EQ-5D version (EQ-5D-5L) essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Visual Analog Scale (Pain) | 6 weeks
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Hospital Anxiety and Depression Scale (HADS, Anxiety and depression) | 6 weeks
  The HADS scale is a questionnaire commonly used to assess patient/client levels of Anxiety and Depression. HADS is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity of anxiety and depression disorders in clients with illness and the general population.The two sub-scales, anxiety and depression, have been found to be independent measures. In its current form the HADS is now divided into four stages:
  Scores of:
  0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Caner KARARTI, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhn JE, Dunn WR, Sanders R, An Q, Baumgarten KM, Bishop JY, Brophy RH, Carey JL, Holloway BG, Jones GL, Ma CB, Marx RG, McCarty EC, Poddar SK, Smith MV, Spencer EE, Vidal AF, Wolf BR, Wright RW; MOON Shoulder Group. Effectiveness of physical therapy in treating atraumatic full-thickness rotator cuff tears: a multicenter prospective cohort study. J Shoulder Elbow Surg. 2013 Oct;22(10):1371-9. doi: 10.1016/j.jse.2013.01.026. Epub 2013 Mar 27. PMID 23540577
- [Background] Ranebo MC, Bjornsson Hallgren HC, Holmgren T, Adolfsson LE. Surgery and physiotherapy were both successful in the treatment of small, acute, traumatic rotator cuff tears: a prospective randomized trial. J Shoulder Elbow Surg. 2020 Mar;29(3):459-470. doi: 10.1016/j.jse.2019.10.013. Epub 2020 Jan 7. PMID 31924516
- [Background] Kukkonen J, Joukainen A, Lehtinen J, Mattila KT, Tuominen EK, Kauko T, Aarimaa V. Treatment of Nontraumatic Rotator Cuff Tears: A Randomized Controlled Trial with Two Years of Clinical and Imaging Follow-up. J Bone Joint Surg Am. 2015 Nov 4;97(21):1729-37. doi: 10.2106/JBJS.N.01051. PMID 26537160
- [Background] Awotidebe AW, Inglis-Jassiem G, Young T. Low-level laser therapy and exercise for patients with shoulder disorders in physiotherapy practice (a systematic review protocol). Syst Rev. 2015 Apr 30;4:60. doi: 10.1186/s13643-015-0050-2. PMID 25925768
- [Background] Haslerud S, Magnussen LH, Joensen J, Lopes-Martins RA, Bjordal JM. The efficacy of low-level laser therapy for shoulder tendinopathy: a systematic review and meta-analysis of randomized controlled trials. Physiother Res Int. 2015 Jun;20(2):108-25. doi: 10.1002/pri.1606. Epub 2014 Dec 2. PMID 25450903